CLINICAL TRIAL: NCT02620761
Title: Fenoldopam to Prevent Renal Dysfunction in Indomethacin Treated Preterm Infants
Acronym: Fenaki
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inability to recruit patients
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jeffrey Segar, Professor of Pediatrics, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DK113073-01A1
Record Dates: First submitted 2015-10-27; First posted 2015-12-03 (Estimated); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Patent Ductus Arteriosus (PDA); Acute Kidney Injury (AKI)
MeSH Terms: conditions — Ductus Arteriosus, Patent; Acute Kidney Injury | interventions — Fenoldopam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Infants in the Placebo arm will receive 0.9% sodium chloride (0.1 ml/hr). If, after 6 hrs there is not a clinically concerning decrease in blood pressure, as determined by attending physician, the rate of infusion (in this arm the placebo) will be increased to 0.2 ml/kg/hr. This rate will be continued throughout the remainder of the study.
  Interventions: Drug: 0.9%NS
- Fenoldopam (Experimental): Infants in the experimental arm will receive fenoldopam (60 ug/ml; 0.1 ml/hr to provide 0.1ug/kg/min). If, after 6 hrs there is not a clinically concerning decrease in blood pressure, as determined by attending physician, the rate of infusion will be increased to 0.2 ml/kg/hr (0.2 ug/kg/min for infants receiving fenoldopam). This rate will be continued throughout the remainder of the study.
  Interventions: Drug: Fenoldopam

INTERVENTIONS:
Drug: Fenoldopam — Randomized to receive Fenoldopam or 0.9%NS
  Arms: Fenoldopam
Drug: 0.9%NS — Randomized to receive Fenoldopam or 0.9%NS
  Other Names: normal saline
  Arms: Control

SUMMARY:
The investigators will conduct a prospective, blinded, randomized, placebo-controlled trial with a sample size of 20 patients in each of the two arms (fenoldopam vs placebo) based upon a difference in serum creatinine by one standard deviation. Fluid and salt intake will be held constant within clinical parameters and carefully measured. Fenoldopam will be started at 0.1 ug/kg/min. If, after 6 hrs there is no decrease in blood pressure, the dose will be increased to 0.2 ug/kg/min. This dose will be continued throughout the remainder of the study. A study of pediatric patients previously provided to the FDA showed no hypotension at a dose of 0.2 ug/kg/min. Fenoldopam will be started 12 hrs before the first dose of indomethacin and discontinued 12 hrs after the 3rd dose of indomethacin. Study samples will include both blood and urine. The primary outcome will be a reduction in renal dysfunction, as determined by creatinine and urine output over the course of treatment. Additional outcomes will include determination of known and novel metabolomic urine markers of renal dysfunction.

DETAILED DESCRIPTION:
Hypotheses

* The investigators primary hypothesis is that fenoldopam reduces renal dysfunction associated with indomethacin administration for closure of patent ductus arteriosus in preterm infants. A secondary endpoint or measured outcome will be the determination of fenoldopam pharmacokinetics in the premature population. Lastly, the investigators hypothesize that urine and serum acute kidney injury (AKI) biomarkers will be superior to contemporary neonatal AKI definitions in their ability to identify renal injury.

Specific Aims

* Evaluate the effect of fenoldopam on renal function in preterm infants administered indomethacin
* Determination of fenoldopam pharmacokinetic and pharmacodynamic profiles in preterm infants
* Define whether newly identified biomarkers of renal dysfunction are more sensitive markers of renal dysfunction following indomethacin than traditional markers including urine output and serum creatinine.

Study design

* The study will be a prospective, blinded, randomized, placebo controlled trial. Fenoldopam will be started at 0.1 ug/kg/min. If, after 6 hrs there is no decrease in blood pressure, the dose will be increased to 0.2 ug/kg/min and continued throughout the remainder of the study. The previous study in pediatric patients showed no hypotension at a dose of 0.2 ug/kg/min. Fenoldopam will be started 12 hrs before the first dose of indomethacin and discontinued 12 hrs after the 3rd dose of indomethacin.

Describe study population or sample material

* preterm infants born at less than or equal to 28 weeks gestation with patent ductus arteriosus in whom attempted medical closure with indomethacin is indicated as decided upon by the attending physician Sample size/power of primary endpoint
* Sample size is 20 patients in each of the two arms (fenoldopam vs placebo) based upon an improvement in serum creatinine by one standard deviation.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age at birth 23 0/7 to 27 6/7 weeks by best obstetrical dating
2. No previous exposure to indomethacin
3. Clinical determination to use indomethacin to attempt closure of PDA
4. No known congenital abnormalities involving the kidneys, heart or lungs
5. No preexisting renal dysfunction, defined as serum creatinine > 1.0 mg/dl, or urine output <1.0 ml/kg/hour over the previous 24 hours.

Exclusion Criteria:

1. Enrollment in concurrent study in which interventions may contribute confounding variables or have competing outcomes
2. Infants with antenatally or postnatally diagnosed renal or urinary tract abnormalities
3. Infants with umbilical cord or infant blood pH below 7.0 at any time before enrollment
4. Attending physician unwilling to have infant participate in study
5. Absence of informed consent

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Segar, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Fenoldopam
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No analysis performed as only a single patient was enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Fenoldopam | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: weeks gestation] | 25 (0) |  | 25 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Urine Output (ml/kg/hr)
Description: Urine will be collected and measured in 6 hour increments beginning 6 hours prior to starting fenoldopam or placebo infusion. The first dose of indomethacin will be given 12 hours after starting fenoldopam or placebo. Two additional doses of indomethacin will be given 12 hours apart. Urine will continue to be collected and volume measured in 6 hour increments up to 24 hrs after the last dose of indomethacin. To summarize, urine will be collected and measured from time -6 hours to 0 hours. Fenoldapam or placebo will be initiated at time 0 hrs, indomethacin given at time 12, 24 and 36 hours, and urine collected and measured to time 60 hours.
Time Frame: 66 hrs - from 6 hrs before beginning of fenoldopam or placebo infusion up to 24 hours after the last dose of indomethacin
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Serum Levels of Fenoldopam During Infusion of the Drug and Following Discontinuation of the Drug Will be Measured by Liquid Chromatography and Mass Spectroscopy.
Description: Blood samples for determination of serum fenoldopam levels will be obtained immediately prior to starting the infusion of fenoldopam (time 0 hour), continue through the 48 hour period of fenoldopam infusion and continue for an additional 12 hours after stopping the fenoldopam infusion.
Time Frame: 60 hours
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Levels of Serum Albumin (mg/dl)
Description: Period from just prior to first dose of indomethacin (time point 12 hours) to 24 hours beyond last dose of indomethacin ( which is time point 60 hours). Thus, this aspect of study takes place between time point 12 hr and time point 60 hr, which is a 48 hour period
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Changes in Serum Creatinine (mg/dl)
Description: Serum creatinine will be measured immediately prior to first dose of indomethacin, immediately prior to the third dose of indomethacin (24 hr later) and 24 hours after the third dose of indomethacin
Time Frame: 48 hours
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Serum Levels of Fenoldopam Will be Related the Changes in Urine Volume
Description: We will relate serum levels of fenoldopam to changes in urine volume over the duration of time of fenoldopam infusion and after discontinuation of infusion. This constitutes part of the pharmacodynamic analysis
Time Frame: 60 hours
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Serum Levels of Fenoldopam Will be Related to Absolute and Relative Changes in Serum Creatinine
Description: We will relate serum levels of fenoldopam to serum creatinine values over the duration of time of fenoldopam infusion and after discontinuation of infusion. This constitutes part of the pharmacodynamic analysis
Time Frame: 60 hours
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Change in Levels of Serum Beta 2 Macroglobulin (mcg/ml)
Description: as for outcome 3
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Change in Levels of Serum Cystatin C (mcg/ml)
Description: as for outcome 3
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Change in Levels of Serum Epidermal Growth Factor (EGF) (ng/ml)
Description: as for outcome 3
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Change in Levels of Serum Osteopontin (ng/ml)
Description: as for outcome 3
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Change in Levels of Serum Uromodulin (mg/dl)
Description: as for outcome 3
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Change in Level of Urine Albumin (mg/dl)
Description: as for outcome 3
Time Frame: 48 hr
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Change in Level of Urine Beta 2 Macroglobulin (mcg/ml)
Description: as for outcome 3
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Change in Level of Urine Cystatin C (mcg/ml)
Description: as for outcome 3
Time Frame: 48 hr
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Change in Levels of Urine Epidermal Growth Factor (EGF) (ng/ml)
Description: as for outcome 3
Time Frame: 48 hr
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Change in Levels of Urine Osteopontin (ng/ml)
Description: as for outcome 3
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Change in Levels of Urine Uromodulin (mg/dl)
Description: as for outcome 3
Time Frame: 48 hrs
Population: No analysis performed as only single patient was enrolled
Arm/Group | Control | Fenoldopam
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Two weeks
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events as per clinicaltrial.gov definitions
Arm/Group | Control | Fenoldopam
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT02620761/Prot_SAP_000.pdf